CLINICAL TRIAL: NCT04957771
Title: Effect of Standardized Exercise on Cardiopulmonary Function in Patients With Permanent Pacemaker Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LM2019185
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2019-08

CONDITIONS: Pacemaker DDD; Cardiopulmonary Endurance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular exercise group (Experimental)
  Interventions: Other: Supervise and guide regular exercise
- non-regurlar exercise group (No Intervention)

INTERVENTIONS:
Other: Supervise and guide regular exercise — Aerobic exercise, evaluated by cardiopulmonary exercise test, 3-5 times a week
  Arms: Regular exercise group

SUMMARY:
The purpose of this study is to observe the changes of cardiopulmonary endurance in patients with pacemaker implantation after long-term exercise, to explore the significance of exercise on patients with pacemaker implantation, and to analyze the difference of the effect of exercise on cardiopulmonary endurance in patients with normal LVEF of different pacing ratios

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old patients with pacemaker implantation for the first time,
* 3-6 months after operation
* stable condition,
* independent walking ability.

Exclusion Criteria:

* Cognitive impairment;
* ICD, CRT / Crtd implanted,
* patients with neurogenic syncope;
* Atrial tachycardia, atrial fibrillation,
* NYHA class II or above,
* difficult to control hypertension;
* Musculoskeletal disease limiting activity
* nervous system disease,
* severe respiratory disease,
* Patients with acute inflammation,
* cancer and other diseases uncontrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Parameters related to exercise cardiopulmonary assessment | followed up for one year
  VO2peak

CONTACTS AND LOCATIONS:
Overall Officials: lijie sun, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: Undecided